CLINICAL TRIAL: NCT00088153
Title: Effects of Anorexia Nervosa on Peak Bone Mass
Brief Title: Effects of Anorexia Nervosa on Bone Mass in Adolescents
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Madhusmita Misra, Chief, Pediatric Endocrinology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK062249; R01DK062249 (NIH)
Record Dates: First submitted 2004-07-20; First posted 2004-07-21 (Estimated); Results first posted 2011-10-10 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Amenorrhea; Bone Mass; Growth hormone
MeSH Terms: conditions — Anorexia Nervosa; Amenorrhea | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiologic estrogen replacement (Experimental): Mature girls with anorexia nervosa (AN) (bone age 15 or greater): Transdermal estradiol (100 mcg) with cyclic progesterone (days 1-10 of each month).
  Immature girls with AN (bone age less than 15 years): Ethinyl estradiol (3.75 mcg daily for the first 6 months, 7.5 mcg daily for the next 6 months, and 11.25 mcg daily for the final 6 months of the study
  Interventions: Drug: Physiologic Estrogen/progesterone
- Placebo (Placebo Comparator): Placebo patches or pills
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Physiologic Estrogen/progesterone — Vivelle Dot patch 100 mcg twice weekly; Provera 2.5 mg daily for the first 10 days of the month
  Other Names: Bone age >=15: Vivelle Dot patch with cyclic Provera
  Arms: Physiologic estrogen replacement
Other: Placebo — Placebo patches twice weekly; Placebo pills daily for the first 10 days of every month
  Arms: Placebo

SUMMARY:
This study is to determine the effects of anorexia nervosa on bone mass and hormone levels in adolescents. Whether administration of estrogen, a normal hormone present during puberty, can help maintain bone development in girls with anorexia nervosa will be determined.

DETAILED DESCRIPTION:
Adolescence is a critical time for bone mineral accretion as between 60-90% of peak bone mass is established during this period, and peak bone mass is a major determinant of bone density and osteoporosis risk during adulthood. Anorexia nervosa (AN) is the third most common chronic illness among adolescent girls, with a prevalence of 0.2-1.0%. Therefore, AN occurs at a time during which patients are the most vulnerable to disruption of bone mineral accretion. Osteopenia is a major co-morbid complication of AN in 50-75% of female adolescents and adult women with this eating disorder. Women with the onset of the disorder during adolescence have more severe osteopenia than women with onset during adulthood. Little is known about the pathogenesis of osteopenia in this adolescent population and there are no established therapies. Improved understanding of bone mineral metabolism and factors which predict recovery of bone mineral accretion are critical in the development of therapeutic strategies to preserve and maximize bone mass in girls with the onset of AN during adolescence. Estrogen is known to be a critical factor in the development of peak bone mass. Although AN is associated with profound estrogen deficiency, there are no controlled studies investigating the effects of estrogen administration in this population.

This research proposal will address critical unanswered questions regarding bone abnormalities in adolescents with anorexia nervosa. Defining changes in bone formation with weight recuperation and hormonal variables would provide insight into the factors essential for bone mineral accretion during adolescence, as well as those that predict recovery. Determination of dose-dependent estrogen effects in this population will be key in targeting interventions during the time of active disease, with the long-term goal of preserving peak bone mass accretion in this vulnerable group of patients. Data obtained from women with post-menopausal osteoporosis or from women with AN cannot be extrapolated to adolescent patients who are in an active period of bone growth and mineralization as well as remodeling. Given the increasing prevalence of AN and its profound consequences on bone health, these studies will provide much needed data to enable treatment strategies for this severe co-morbid disease.

ELIGIBILITY:
Inclusion Criteria:

* Females Only with Anorexia Nervosa and Amenorrhea 12-18 years
* Normal-weight girls 12-18 years with no past or present history of an eating disorder

Exclusion Criteria:

* Diseases affecting bone metabolism (including untreated thyroid disease, premature ovarian failure, diabetes, cancer, pituitary, renal disease or bone fracture within the past six months)
* Use of prescription medications affecting bone metabolism within three months
* Suicidality
* Psychosis
* Substance abuse
* Hematocrit <30 %
* Potassium <3.0 mmol/L
* Glucose <50 mg/dl.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2003-07; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhusmita Misra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Misra M, Katzman D, Miller KK, Mendes N, Snelgrove D, Russell M, Goldstein MA, Ebrahimi S, Clauss L, Weigel T, Mickley D, Schoenfeld DA, Herzog DB, Klibanski A. Physiologic estrogen replacement increases bone density in adolescent girls with anorexia nervosa. J Bone Miner Res. 2011 Oct;26(10):2430-8. doi: 10.1002/jbmr.447. PMID 21698665
- [Derived] Misra M, Katzman DK, Estella NM, Eddy KT, Weigel T, Goldstein MA, Miller KK, Klibanski A. Impact of physiologic estrogen replacement on anxiety symptoms, body shape perception, and eating attitudes in adolescent girls with anorexia nervosa: data from a randomized controlled trial. J Clin Psychiatry. 2013 Aug;74(8):e765-71. doi: 10.4088/JCP.13m08365. PMID 24021517
- [Derived] Faje AT, Fazeli PK, Katzman DK, Miller KK, Breggia A, Rosen CJ, Mendes N, Klibanski A, Misra M. Sclerostin levels and bone turnover markers in adolescents with anorexia nervosa and healthy adolescent girls. Bone. 2012 Sep;51(3):474-9. doi: 10.1016/j.bone.2012.06.006. Epub 2012 Jun 15. PMID 22728230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period of recruitment: 2003-2009. Location: Massachusetts General Hospital (Boston) and Hospital for Sick Children (Toronto).
  We screened 150 girls with anorexia nervosa (AN) (110 at MGH and 40 at SickKids) and 88 normal-weight controls 12-18 years. Following the screen, 110 AN and 40 controls were enrolled for the prospective study.
Pre-assignment Details: Reasons for enrolled participants being excluded from the trial before assignment to groups primarily included identification of exclusion criteria, loss of interest on the part of the participant, and loss to follow-up.
Groups:
- Physiologic Estrogen Replacement: Mature girls with anorexia nervosa (bone age 15 or greater): Transdermal estradiol (100 mcg) with cyclic progesterone (days 1-10 of each month).
  Immature girls with anorexia nervosa (bone age less than 15 years): Ethinyl estradiol (3.75 mcg daily for the first 6 months, 7.5 mcg daily for the next 6 months, and 11.25 mcg daily for the final 6 months of the study
- Placebo: Mature girls with anorexia nervosa with a bone age of 15 years of greater: Placebo patches; Immature girls with anorexia nervosa with a bone age of less than 15 years: Placebo pills
Period: Overall Study
Arm/Group | Physiologic Estrogen Replacement | Placebo
Started | 55 | 55
Completed | 31 | 30
Not Completed | 24 | 25
Not completed — Physician Decision | 3 | 3
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Lost to Follow-up | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physiologic Estrogen Replacement | Placebo | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 55 | 55 | 110
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (1.6) | 16.3 (1.6) | 16.5 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Spine Bone Density Over the Study Duration (18 Months)
Description: Bone density at the spine (lumbar 1-4 vertebrae) was measured using dual energy x-ray absorptiometry (DXA) at baseline, 6 months, 12 months and 18 months.
  The primary outcome was the percent change in bone density at the spine from baseline to 18 months. Areal bone density is measured as g/cm2. The unit of measure for the percent change in bone density is 'percent' Percent change in bone density= [[Bone density at 18 months- Bone density at baseline)*100/Bone density at baseline]%
Time Frame: Baseline and 18 months
Population: The number of participants was determined using power calculations based on preliminary data. For our primary longitudinal analysis, bone mineral density (BMD) changes were analyzed using a mixed model analysis of variance (intent-to-treat model). For secondary analysis, we examined BMD changes after controlling for age and weight changes.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Physiologic Estrogen Replacement: Mature girls with anorexia nervosa (AN) (bone age ≥15 years) randomized this arm received transdermal 17-β estradiol (100 mcg patch applied twice weekly) continuously over the study duration. Girls randomized to the active estradiol patch also received medroxyprogesterone 2.5 mg daily for 10 days each month. Immature girls with AN (bone age<15 years, N=14) randomized to this arm received escalating doses of oral ethinyl estradiol (3.75 mcg daily for the first 6 months, 7.5 mcg daily for the second 6 months, and 11.25 mcg daily for the last 6 months). All subjects were given 1200 mg calcium carbonate and 400 IU vitamin D daily.
- Placebo: Mature girls with anorexia nervosa (AN) randomized to this arm received placebo patches and cyclic placebo pills.
  Immature girls with AN randomized to this arm received placebo pills. All subjects received supplemental calcium (1200 mg) and vitamin D (400 IU) daily
Arm/Group | Physiologic Estrogen Replacement | Placebo
Number analyzed (Participants) | 55 | 55
Percent change | 2.6 (1.0) | 0.3 (0.1)
Statistical Analysis 1: Comparison: Physiologic Estrogen Replacement vs Placebo; Power analysis: We have previously demonstrated that normal female adolescents gain bone density at the rate of 0.039 +/- 0.0507 per year. The pooled SD in that study was 0.046. Based on these data, with a sample size of 110 girls with anorexia nervosa (AN), half of whom are randomized to receive estrogen and half placebo (with a 10% drop-out rate), there will be an 80% chance that we will detect an increase in bone density to 75% of normal in the girls who receive estrogen; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — After controlling for baseline age and weight changes; We also used a mixed model analysis of variance (PROC MIXED), to analyze longitudinal data

2. Secondary Outcome: Change in N-terminal Propeptide of Type 1 Procollagen (P1NP) Over the Study Duration (18 Months)
Description: P1NP is a surrogate marker of bone formation that is measured in serum. P1NP levels were measured at baseline, 6, 12 and 18 months.
  A secondary outcome was the change in P1NP levels from baseline to 18 months: [P1NP at 18 months - P1NP at baseline). The unit is ng/ml
Time Frame: Baseline and 18 months
Population: The number of participants was determined based on our preliminary data. This analysis was based on completers only.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Physiologic Estrogen Replacement | Placebo
Number analyzed (Participants) | 55 | 55
ng/ml | -2.9 (22.5) | -10.9 (27.0)
Statistical Analysis 1: Comparison: Physiologic Estrogen Replacement vs Placebo; The null hypothesis was that there would be no differences between the groups for changes in P1NP levels over time; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

3. Primary Outcome: Change in Spine Bone Mineral Density Z-scores Over the Study Duration (18 Months)
Description: Bone density at the spine (lumbar 1-4 vertebrae) was measured using dual energy x-ray absorptiometry (DXA) at baseline, 6 months, 12 months and 18 months.
  The other primary outcome was the change in spine bone density Z-score from baseline to 18 months. The bone density Z-score is a standard deviation score that compares one's bone density to the mean for age and gender, and the Z-score, therefore, does not have any units. It is simply referred to as a Z-score. Change in bone density Z-score= [Bone density Z-score at 18 months- Bone density Z-score at baseline]
Time Frame: Baseline and 18 months
Measure: Mean (Standard Deviation); unit: Z -scores
Arm/Group | Physiologic Estrogen Replacement | Placebo
Number analyzed (Participants) | 55 | 55
Z -scores | -0.026 (0.078) | -0.236 (0.091)
Statistical Analysis 1: Comparison: Physiologic Estrogen Replacement vs Placebo; The null hypothesis was that the groups would not differ for changes in spine bone density z-scores over the study duration; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The p value was adjusted for age and weight changes

ADVERSE EVENTS:
Time Frame: 18 months for each subject(AN E+ versus AN E-)
Arm/Group | Physiologic Estrogen Replacement | Placebo
Serious Adverse Events (participants affected / at risk) | 12/55 | 16/55
Other Adverse Events (participants affected / at risk) | 18/55 | 20/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physiologic Estrogen Replacement (N=55) | Placebo (N=55)
Hospitalizations for low weight and/or bradycardia (General disorders) | 12 (12) | 16 (16)
Increased vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erythema at patch application site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pregnancy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physiologic Estrogen Replacement (N=55) | Placebo (N=55)
Nausea/vomiting (Gastrointestinal disorders) | 14 (14) | 8 (8)
Dizziness (Vascular disorders) | 6 (6) | 10 (10)
Headaches (Nervous system disorders) | 10 (10) | 14 (14)
Bloating (Gastrointestinal disorders) | 18 (18) | 16 (16)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4)
Breast tenderness (Reproductive system and breast disorders) | 14 (14) | 9 (9)
Increased vaginal discharge (Reproductive system and breast disorders) | 13 (13) | 9 (9)
Increased uterine bleeding (Reproductive system and breast disorders) | 13 (13) | 9 (9)
Irritation from contact lenses (Eye disorders) | 2 (2) | 6 (6)
Perceived increase in facial hair (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Perceived loss of scalp hair (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5)
Worsening depression (Psychiatric disorders) | 3 (3) | 5 (5)
Erythema at patch application site (Skin and subcutaneous tissue disorders) | 17 (17) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No